CLINICAL TRIAL: NCT03624920
Title: Safety and Efficacy of THN102 in Patients With Parkinson's Disease and Excessive Daytime Sleepiness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theranexus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: THN102-202
Record Dates: First submitted 2018-07-10; First posted 2018-08-10 (Actual); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Complete 3 way-Crossover
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- THN102 Dosage A (Placebo Comparator): THN102 Dosage A is a Placebo
  Interventions: Drug: THN102 Dosage A
- THN102 Dosage B (Experimental): THN102 Dosage B : 200 mg/2 mg THN102 is a combination of modafinil 100mg and flecainide 1 mg daily dosage is 200 mg of modafinil and 2 mg of flecainide
  Interventions: Drug: THN102 Dosage B
- THN102 Dosage C (Experimental): THN102 Dosage C : 200 mg/18 mg THN102 is a combination of modafinil 100mg and flecainide 9 mg daily dosage is 200 mg of modafinil and 18 mg of flecainide
  Interventions: Drug: THN102 Dosage C

INTERVENTIONS:
Drug: THN102 Dosage A — THN102 Dosages A: placebo
  Other Names: Placebo
  Arms: THN102 Dosage A
Drug: THN102 Dosage B — THN102 Dosage B : 200mg/2mg
  Other Names: Dosage B
  Arms: THN102 Dosage B
Drug: THN102 Dosage C — THN102 Dosage C: 200mg/18mg
  Other Names: Dosage C
  Arms: THN102 Dosage C

SUMMARY:
This is a randomized, placebo-controlled, 3-way cross-over phase IIa trial comparing two dose levels of THN102 to placebo in patients suffering from Parkinson's disease associated with excessive daytime sleepiness.

DETAILED DESCRIPTION:
The treatment duration is 2 weeks per period. Each treatment period is followed by a one-week washout period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of idiopathic Parkinson's disease as defined by the Movement Disorders Society (MDS).
* Subjects with Hoehn and Yahr scale score ≤ 4.
* Body mass index > 18 kg/m2 and < 35 kg/m2.
* Subjects should have a complaint of daytime sleepiness impacting their quality of life and/or daytime functioning (e.g. falling asleep while reading or watching television, while eating or talking with other people).
* Epworth Sleepiness Scale (ESS) score ≥ 14.

Exclusion Criteria:

* Subjects with known or with a suspected sleep apnea syndrome or who have any other cause of excessive daytime sleepiness, such as shift work sleep disorder.
* Psychiatric and neurological disorders (other than Parkinson's disease),
* Cardiovascular disorders such as - but not limited to
* Uncontrolled moderate to severe hypertension
* History or current diagnosis of electrocardiogram (ECG) abnormalities indicating significant risk of safety for patients participating in the study
* Recent myocardial infarction
* Stable or unstable angina pectoris
* Cardiac insufficiency or history of heart failure
* Previous history of cardiac valvular surgery
* Subjects with current impulse control disorder.
* Subjects showing dementia or with MoCA < 23.
* Subjects with current suicidal risk
* Current or recent (within one year) history of substance abuse or dependence disorder
* Other active clinically significant illness
* Subjects with hepatic or renal impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Corvol, Prof, Study Chair — Hôpital La Pitié-Salpêtrière, 75651 Paris, France, Tel. +33 1 42 16 57 66, mail: jean-christophe.corvol@aphp.fr
Locations (34):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - MGH Neurological Clinical Research Institute, Boston, Massachusetts
  - Houston Methodist Hospital, Houston, Texas
- Czechia (8):
  - I. neurologická klinika Fakultní nemocnice u sv. Anny, Brno
  - Neurologická klinika Fakultní nemocnice Hradec Králové, Hradec Králové
  - Neurologická klinika Fakultní nemocnice Ostrava, Ostrava Poruba
  - Neurologická klinika 1.LF UK a VFN v Praze, Prague
  - NEURO - Praha, s.r.o., Prague
  - Axon Clinical, s.r.o., Prague
  - Neurologické oddělení Nemocnice Na Homolce, Prague
  - Institut neuropsychiatrické péče, Prague
- France (7):
  - Hôpital NEurologique Pierre Wertheimer, Bron
  - CHRU Hopital Salengro, Lille
  - CHU de la Timone Service de Neuro et pathologie du mouvement, Marseille
  - CHRU Guy de Chauliac, Montpellier
  - ICM Centre d'Investigation Clinique Hôpital Pitié Salpêtrière, Paris
  - CHU Charles Nicolle, Rouen
  - CHU Purpan CIC Hall D 2eme etage, Toulouse
- Germany (9):
  - Praxis Dr. Safavi, Neuroakademie Alzenau, Alzenau in Unterfranken
  - Charité - Universitätsmedizin Berlin, Klinik für Neurologie, Campus Benjamin Franklin, Berlin
  - Neurologische Praxis Dipl. med. Christian Oehlwein, Gera
  - Pharmakologisches Studienzentrum Chemnitz, Mittweida
  - Technische Universität München, Klinikum rechts der Isar, Neurologische Klinik und Poliklinik, Neuro-Kopf-Zentrum, München
  - Praxis Dr. med. Arnfin Bergmann, Neuburg am Inn
  - Neurozentrum Sophienstrasse, Stuttgart
  - NeuroPoint, Ulm
  - Gemeinschaftspraxis Dr. med. Joachim Springub / Wolfgang Schwarz, Studienzentrum Nord-West, *ausgelagerte Praxisräume:, Westerstede
- Hungary (7):
  - Nyírő Gyula Országos Pszichiátriai és Addiktológiai Intézet, Neurológiai Osztály, Budapest
  - Észak-Közép-budai Centrum, Budapest
  - Debreceni Egyetem Kenézy Gyula Egyetemi Kórház Neurológiai Osztály, Debrecen
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktató Kórház, Stroke, Vascularis és Általános Neurológiai és Toxikológiai Osztály, Miskolc
  - PTE KK Neurológiai Klinika, Pécs
  - Szegedi Tudományegyetem ÁOK Szent-Györgyi Albert Klinikai Központ Neurológiai Klinika, Szeged
  - Theranexus Investigational site, Szeged

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 105 patients were screened and 77 were randomized and allowed to start the medications periods.
Groups:
- Sequence ABC; Sequence BCA; Sequence CAB; Sequence ACB; Sequence CBA; Sequence BAC: A : 2 weeks under Placebo
  B : 2 weeks under THN102 200/2 (200mg modafinil and 2 mg of flecainide per os daily)
  C : 2 weeks under THN102 200/18 (200mg modafinil and 18 mg of flecainide per os daily)
Period: Overall Study
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB | Sequence ACB | Sequence CBA | Sequence BAC
Started | 14 | 14 | 13 | 13 | 11 | 12
Completed | 13 | 12 | 12 | 12 | 7 | 11
Not Completed | 1 | 2 | 1 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Population: mITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB | Sequence ACB | Sequence CBA | Sequence BAC | Total
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 9 | 11 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 7 | 9 | 4 | 3 | 34
  >=65 years | 8 | 7 | 6 | 4 | 5 | 8 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 9 | 9 | 7 | 9 | 48
  Male | 5 | 7 | 4 | 4 | 2 | 2 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : White | 13 | 13 | 12 | 13 | 9 | 11 | 71
  Race Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Ethnicity : Not hispanic or latino | 13 | 12 | 12 | 13 | 8 | 11 | 69
  Ethnicity : Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Ethnicity : not reported | 0 | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety Adverse Events
Description: Number of participants with spontaneously reported treatment-related adverse events
Time Frame: 2 weeks
Population: Overall number of participant reported corresponds to the safety set population of the clinical report
Measure: Number; unit: participants
Groups:
- Placebo: THN102 Placebo (Dosage A)
- THN102 200/2: THN102 200 mg/2 mg (Dosage B)
- THN102 200/18: THN102 200 mg/18 mg (Dosage C)
Arm/Group | Placebo | THN102 200/2 | THN102 200/18
Number analyzed (Participants) | 68 | 72 | 73
participants
  Subjects with at least one TEAE leading to death | 0 | 0 | 0
  Subject with at least one serious TEAE | 0 | 0 | 1
  Subjects with at least one related serious TEAE | 0 | 0 | 0
  Subjects with at least one TEAE | 19 | 23 | 29
  Subjects with at least one related TEAE | 5 | 11 | 18
  Subjects with at least one TEAE leading to discont | 0 | 3 | 3
  Subjects with at least one related TEAE leading to | 0 | 2 | 3
  Subjects with at least one serious TEAE leading to | 0 | 0 | 0

2. Secondary Outcome: Epworth Sleeping Scale (ESS)
Description: Range of the scale : 0 to 24. A low score indicates a good outcome. Results shown are corresponding to a change from baseline of the ESS score.
Time Frame: 2 weeks
Population: modified intent to treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | THN102 200/2 | THN102 200/18
Number analyzed (Participants) | 68 | 70 | 72
score on a scale | -2.4422 (0.5117) | -3.8417 (0.5086) | -3.1850 (0.4982)

3. Secondary Outcome: Psychomotor Vigilance Test (PVT) : Reaction Time (Miliseconds) Change From Baseline
Description: PVT measures reaction time in milliseconds. The results below are corresponding to the reaction time change from baseline.
Time Frame: 2 weeks
Population: PVT full analysis set
Measure: Least Squares Mean (Standard Error); unit: millisecond (msec)
Arm/Group | Placebo | THN102 200/2 | THN102 200/18
Number analyzed (Participants) | 68 | 70 | 72
millisecond (msec) | -21.2201 (10.0565) | -24.1089 (9.9393) | -19.6450 (9.8847)

4. Secondary Outcome: Montreal Cognitive Assessment Battery (MoCA)
Description: MoCA score reflects the cognitive capacities of a person. Range of the total score of 10 test items: 0 to 30 points. A high score indicates good cognitive functioning. A score of 26 and above is considered normal.
  The results below are shown as change from baseline of the MoCA score.
Time Frame: 2 weeks
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | THN102 200/2 | THN102 200/18
Number analyzed (Participants) | 68 | 70 | 72
score on a scale | 0.2240 (0.1935) | 0.03267 (0.1923) | 0.4251 (0.1900)

5. Secondary Outcome: Efficacy in Improving Sleepiness (ESS). Responders Rate, Change From Baseline
Description: ESS score responder rate, defined as the proportion of subjects with at least 25% ESS improvement from baseline, at the end of each treatment period
Time Frame: 2 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | THN102 200/2 | THN102 200/18
Number analyzed (Participants) | 68 | 69 | 71
Participants | 19 | 28 | 25

6. Secondary Outcome: Efficacy in Improving Sleepiness (ESS). Patients in Remission, Change From Baseline
Description: Number of patients in remission (=without residual sleepiness), i.e. ESS < 11 at the end of each treatment period
Time Frame: 2 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | THN102 200/2 | THN102 200/18
Number analyzed (Participants) | 68 | 69 | 71
Participants | 11 | 19 | 18

ADVERSE EVENTS:
Time Frame: AE collection through study duration, starts with screening until follow up visit (last phone call), a total of 13 weeks.
Description: Listing of AEs reported are corresponding to TEAEs (treatment emergent adverse event) collected from randomization to last visit
Groups:
- THN102 Placebo: THN102 Placebo (Dosage A)
Arm/Group | THN102 Placebo | THN102 200/2 | THN102 200/18
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/72 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/72 | 1/73
Other Adverse Events (participants affected / at risk) | 3/68 | 10/72 | 22/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THN102 Placebo (N=68) | THN102 200/2 (N=72) | THN102 200/18 (N=73)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) — wrist contusion and low back pain after fall
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THN102 Placebo (N=68) | THN102 200/2 (N=72) | THN102 200/18 (N=73)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT03624920/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT03624920/SAP_001.pdf